CLINICAL TRIAL: NCT06398951
Title: A Comparison of Conventional High Flow Nasal Cannula vs Two-nare Size High Flow Nasal Cannula: A Randomized Crossover Trial in Extubated Patients
Brief Title: HFNC vs Two Nare HFNC in Extubated Patients
Acronym: HFNC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peninsula Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 87400
Record Dates: First submitted 2024-03-24; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-02

CONDITIONS: Oxygen Deficiency
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two Nare (Duet) high flow nasal cannula (Active Comparator): Recently a new mode of high flow oxygen therapy has presented on the market where the cannula of high flow have different diameters. Left cannula larger in diameter than the right. These two-nare size high flow nasal cannula are capable of delivering gases at a flow rate of 15-60 L/min, similar to the conventional HFNP but the difference in the diameters provide different levels of positive pressure as compared to conventional HFNP. The two nare nasal cannula will be used for 30 minutes to assess the gas exchange, hemodynamic parameters, the tolerance and comfort of the device to the patient.
  Interventions: Device: Two nare high flow nasal cannula
- Conventional High flow nasal cannula (Placebo Comparator): Conventional high flow nasal cannula that has been used for many years will be compared with two-nare high flow nasal cannula. The two nare nasal cannula will be used for 30 minutes to assess the gas exchange, hemodynamic parameters, the tolerance and comfort of the device to the patient.
  Interventions: Device: Two nare high flow nasal cannula

INTERVENTIONS:
Device: Two nare high flow nasal cannula — Recently a new mode of high flow oxygen therapy has presented on the market where the prongs of high flow have different diameters .These two-nare size high flow nasal cannula are capable of delivering gases at a flow rate of 15-50 L/min, similar to the conventional HFNP but the difference in the diameters provide different levels of positive pressure as compared to conventional HFNP.

SUMMARY:
High flow nasal cannula (HFNC) are introduced to clinical practice to improve oxygenation. Our group were the first to report the use of HFNC in extubated patients that showed comparable delivery of oxygen and improved comfort. These HFNC are subsequently shown to be useful in several clinical conditions in critically ill patients including respiratory failure due to hypoxia, hypercapnia (exacerbation of chronic obstructive lung disease), or post-extubation, pre-intubation oxygenation, and others.

Recently a new mode of high flow oxygen therapy has been presented on the market where the prongs of high flow have two different diameters. These two-nare size high flow nasal cannula are capable of delivering gases at a flow rate of 15-50 L/min, similar to the conventional HFNP but the difference in the diameters provide different levels of positive pressure as compared to conventional HFNP. This positive pressure could help in gas exchange of patients who need more oxygen. These devices are approved by the Therapeutic Goods Administration (TGA); the medicine and therapeutic regulatory agency of the Australian Government.

Our aim is to compare the two size nare high flow nasal cannula with conventional high flow nasal cannula in extubated patients in intensive care unit in a randomised crossover trial. The comparison will include arterial blood gasses, physiological data including heart rate, respiratory rate, saturations as well as comfort and tolerance of the patients to two size nare high flow nasal cannuale.

DETAILED DESCRIPTION:
This is a randomised crossover study of ventilated patients suitable for extubation was conducted. Potential patients were clinically assessed for suitability of extubation and arterial blood gasses (ABG) were performed prior to extubation to ensure the patients had optimal gas exchange. If found to be suitable for extubation, patients were extubated and were provided with a high flow blend of oxygen and air by a high flow face mask at a rate of 40 litres per minute delivering an FiO2 to ensure an oxygen saturation of 93% + 1 for 30 minutes. At the end of this 30 minute stabilization, ABG were performed and heart rate, blood pressure, and Glasgow coma score (GCS) were recorded. If the patients remained stable they were randomized to either protocol A (Duet HFNP for 30 minutes followed by conventional HFNP for 30 minutes) or protocol B ( conventional HFNP for 30 minutes followed by Duet HFNP for 30 minutes). During both protocols gas flow rate and FiO2 were maintained at exactly the same settings as used during the stabilization period. Blood gases and other physiological observations (heart rate, blood pressure, and respiratory rate, saturations, GCS, comfort score and tolerance score) were recorded at the end of each protocol. The bed side nurse assessed comfort and tolerance of patients to both the devices by a 5-point Likert scale as shown below. For the purpose of this study only medium size cannulas were used to maintain consistency. Subgroup Comparisions will be performed between those with and without nasogastric tubes and between male and female patients. Randomization is performed using sequentially numbered, sealed, opaque envelope to maintain allocation concealment.

Determine patient's comfort:

Patients provided the comfort for both duet HFNP and conventional HFNP prongs using a 5-point Likert scale;

1. No discomfort,
2. Little bit discomfort,
3. Little more discomfort,
4. Whole lot more discomfort
5. Worst discomfort.

Determine patient's tolerance:

The bedside nurse documented the patient's tolerance using a 5-point Likert scale.

0 Patient never removes the apparatus and does not complain

1. Patient complains about keeping apparatus on
2. Patient request removal of the apparatus
3. Removal of the apparatus by the patient once
4. Removal of multiple times or non-compliance.

ELIGIBILITY:
Inclusion Criteria:

* All intubated patients imminently requiring extubation with family consent for admittance into the trial that meet the follow criteria:
* P/F ratio between > 150 prior to extubation
* Has a functional arterial catheter to allow sample of arterial blood gasses.

Exclusion Criteria:

* Patients being extubated due to withdrawal of therapy Patients being extubated, that are expected to imminently die post extubation P/F Ratio :< 150 Patients extubated on to non-invasive ventilation Patients with known epistaxis or nasal surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Blood gasses (PaO2 in mmHg) | 30 minutes each for a total of one hour.
  To compare if there is difference in PaO2 between two nare and connventional high flow nasal cannula.
Blood gasses (PaCO2 in mmHg) | 30 minutes each for a total of one hour.
  To compare if there is difference in PaCO2 between two nare and connventional high flow nasal cannula.
Blood gasses (SaO2 percentage) | 30 minutes each for a total of one hour.
  To compare if there is difference in SaO2 between two nare and connventional high flow nasal cannula.

SECONDARY OUTCOMES:
blood pressure (mmHg) | 30 minutes each for a total of one hour.
  To compare if there is difference in blood pressure between two nare and connventional high flow nasal cannula.
Respiratory rate (breaths per minute) | 30 minutes each for a total of one hour.
  To compare if there is difference in respiratory rate between two nare and connventional high flow nasal cannula.
Tolerance as assessed by a 5-point Likert scale ranging from 0-4. | 30 minutes each for a total of one hour.
  To compare if there is difference in tolerance assessed by bedside nurse between two nare and connventional high flow nasal cannula.
Comfort as assessed by a 5-point Likert scale ranging from 1-5. | 30 minutes each for a total of one hour.
  To compare if there is difference in comfort as reported by the patient between two nare and connventional high flow nasal cannula.

CONTACTS AND LOCATIONS:
Overall Officials: RAVINDRANATH TIRUVOIPATI, PhD, Principal Investigator — Peninsula Health
Locations (1):
- Frankston Hospital, Frankston, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tiruvoipati R, Reddy MP, Paul E, Gupta S, Subramaniam A, Zhang D, Haji K. A comparison of conventional high-flow nasal cannula vs the duet high-flow nasal cannula in extubated patients: a randomized crossover trial. Eur J Med Res. 2025 Mar 26;30(1):205. doi: 10.1186/s40001-025-02447-0. PMID 40140950